CLINICAL TRIAL: NCT05679427
Title: A Randomised, Prospective, Monoinstitutional Study of Ablative Radiosurgery vs Stereotactic Radiotherapy in 5 Fractions, With Simultaneous Integrated Boost, for the Treatment of Bone Lesions in Oligometastatic Disease
Brief Title: Ablative Radiosurgery vs Stereotactic RT in 5 Fractions With SIB for Oligometastatic Bone Lesions
Acronym: ONES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Nadia Di Muzio, Professor, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONES Trial
Record Dates: First submitted 2022-12-01; First posted 2023-01-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Oligometastatic Disease
Keywords: SBRT; Simultaneous Integrated Boost; Oligometastatic Disease; Bone Metastases
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: The sample size calculation is based on the Kaplan-Meier estimator and uses a log-rank test (Freedman, 1982; Machin et al., 2018). Assuming for the two groups a two-year LRFS of 95% and 85%, respectively, with alpha=0.05 and power of 80%, the total number needed to identify a significant difference between the two curves is 292 (test at 2 queues, 146 patients per group).
  Calculations were performed with software (PASS 2021, v21.0.3). Assuming a 5% dropout, we expect to enroll 15 more patients in total, thus reaching a final number of 307.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Single fraction radiosurgery on bone metastases (21-24Gy x 1 fraction)
  Interventions: Radiation: radiosurgery and stereotactic ablative radiotherapy with simultaneous integrated boost, respectively
- Arm B (Active Comparator): Multi-fractioned stereotactic ablative radiotherapy (5 fractions delivered in 5 consecutive working days) with SIB on bone metastases (5Gy x 5 fractions + SIB up to 40-50Gy)
  Interventions: Radiation: radiosurgery and stereotactic ablative radiotherapy with simultaneous integrated boost, respectively

INTERVENTIONS:
Radiation: radiosurgery and stereotactic ablative radiotherapy with simultaneous integrated boost, respectively — Two protocols of stereotactic ablative radiotherapy, in one vs five fractions ( the later with SIB) are compared

SUMMARY:
This is a randomised prospective monoinstitutional study comparing radiosurgery at a total dose up to 24 Gy to five fraction stereotactic radiotherapy with simultaneous integrated boost (SIB) up to 50 Gy for the treatment of bone metastases in oligometastatic cancer treated with radical intent. At the end of the first 12 months from the start of the study an interim analysis will be performed taking into account all major endpoints for an initial evaluation of the study , with only an observational purpose, without subsequent protocol changes.

DETAILED DESCRIPTION:
The study is interventional, homogeneous (performed in a single institution). Patient recruitment Patients who meet the inclusion criteria will be enrolled during the initial Radiation Oncology examination in our institution or during the multidisciplinary meeting.

Recruitment and selection The patients will be informed of the possibility to participate in the study. I pazienti verranno informati ella possibilità di accedere allo studio. After a careful verification of the inclusion and exclusion criteria, and precise description of the benefits, risks and procedure of the current study, the patient will be asked to sign the informed consent and subsequently randomised.

The following information will be collected for each patient, as is standard practice in our department: demographic data, clinical history, concomitant medical treatments, physical exam, blood exam, tumoral markers, diagnoses CT / Bone scintigraphy/ MRI/ PET and any other staging exam or post tumoral treatment re-evaluation performed.

Randomisation A centralized randomization, with closed envelopes, will be performed by a secretary not involved in the study.

Pre-treatment phase Each patient will undergo the simulation CT, in line with routine clinical practice, with immobilisation devices within 15 (+/- 5) days from the randomisation. The simulation CT will be performed in the Radiotherapy department, the MRI in the Radiology department.

Treatment phase The protocol treatment uses two radiotherapy regimens with ablative doses, which are already included in the daily clinical practice at San Raffaele Scientific Institute and many other national centers equipped with High Technology. The treatment machine will be randomly assigned, depending on the availability of slots for the timing required by the protocol.

The patients will be randomized at a 1:1 ratio between:

* Arm A: radiosurgery ( in one fraction) to the bone metastases ( 21-24 Gy in 1 fraction)
* Arm B: Multifractionated ablative stereotactic radiotherapy (5 fractions, one fraction per day, 5 consecutive weekdays) with SIB to the bone metastases (up to 40-50 Gy).

The treatment should be completed within 1 month from the CT simulation and within 45 (+/- 5) days from randomization (first visit).

Post-treatment phase:

Patients will be evaluated according to departmental clinical practice: at the first visit, at the end of the treatment and at follow-up visits at 3, 6, 12, 18, 24, 36 months from the end of radiotherapy with CT and/or Bone Scan and/or MRI and/or PET/CT based on the treated sites, on the histology of primary tumor, and by means of laboratory exams. Subsequent radiological images of laboratory analyses will be performed at the discretion of the radiation oncologist, based on symptoms or clinical findings. At every visit the anamnesis, physical examination, the CTCAE(Common Terminology Criteria for Adverse Events) toxicity evaluation will be performed and registered, together with any skeletal events, re-irradiation, other systemic therapy lines, or palliative treatment. The patient will fill in the Pain Diary and the quality of life questionnaires (EORTC QLQ-C30, QLQBM22, and EQ-5D-3L). The follow-up visits will be performed in the dedicated rooms of the Radiation Oncology department.

ELIGIBILITY:
Inclusion Criteria:

* Performance status ECOG ≤2
* Life expectancy > 6 months according to Mizumoto criteria*
* Oligometastatic disease (Total number of metastases from 1 to 5: both synchronous and metachronous with maximum involvement of three organs in total - lymph nodes, bones, lungs, liver, adrenal gland, brain- with known histology
* At least one bone metastasis treatable with SABR or SRS
* Each secondary localization (synchronous, metachronous or oligoprogressive) must be treated with radical intent.
* Patients may have received other anticancer treatments (surgery for initial site of disease or other metastases, chemotherapy, radiotherapy for other metastatic sites)

Exclusion Criteria:

* Sites of disease not eligible for stereotactic radiotherapy
* Serious medical comorbidities that preclude RT
* Overlap with a previously treated volume of radiotherapy
* Dimension greater than 5 cm for extra-cranial lesions.
* Size greater than 3 cm for brain lesions
* More than 1 brain metastases
* Clinical or radiological evidence of spinal cord compression or epidural tumor within 2mm of the spinal cord
* Radiological evidence of vertebral body fracture or involvement of more than 40% of the vertebral body
* Radiological evidence of cortical involvement in long bones
* Pregnant or breastfeeding women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2025-11-07 (Estimated); Study Completion 2027-12-07 (Estimated)

PRIMARY OUTCOMES:
Local recurrence-free surival | 3 years from the end of treatment
  evaluation of the impact of stereotactic radiotherapy (one fraction versus fractionated) on local control of disease in terms of local recurrence free survival (LRFS) in patients with oligometastastic disease and at least one bone metastasis.

SECONDARY OUTCOMES:
Acute and late local toxicity | Changes form baseline at 3 years from the end of treatment
  Impact of the two treatments on the local radioinduced toxicity in terms of incidence in skeletal events and acute and late toxicity measured with the Common Terminology Criteria for Adverse Events v5.0 scale
Pain control | Changes form baseline at 3 years from the end of treatment
  Pain control of symptomatic bone lesions measured through the variation of pain diary
Overall survival | 3 years from the end of treatment
  Overall-surival
Cancer Specific Survival | 3 years from the end of treatment
  Cancer Specific Survival
Progression to polymetastatic disease | 3 years from the end of treatment
  Impact of the two treatments on the rate of progression to polymethastatic disease
Adjusted disease-free survival | 3 years from the end of treatment
  defined as the time between the end of radiotherapy and the date of disease progression (local or distant) or the start of therapy (systemic or palliative)
Incidence of Treatment-Emergent Adverse Events as assessed by EORTC-QLQ-C30 | Changes from baseline at 3 years after the treatment
  Quality-of-life assessed by EORTC-QLQ-C30 questionnaire
Incidence of Treatment-Emergent Adverse Events as assessed by EORTC-QLQ-BM22 | Changes from baseline at 3 years after the treatment
  Quality-of-life assessed by EORTC-QLQ-BM22 questionnaire
Satisfaction assessed by EQ-5D-3L | Changes from baseline at 3 years after the treatment
  Quality-of-life assessed by EQ-5D-3L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nadia G Di Muzio, Prof, Principal Investigator — IRCCS San Raffaele, Milan
Locations (1):
- San Raffaele Scientific Institute, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study (anonymized individual participant data) are available on request from the corresponding author to researchers who provide a methodologically sound proposal. Requests made to the corresponding author will be evaluated by the IRCCS San Raffaele Scientific Institute Ethics Committee.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Five years after the end of the study.
Access Criteria: Requests to corresponding author, approved by Ethics Committee

REFERENCES:
- [Background] Hellman S, Weichselbaum RR. Oligometastases. J Clin Oncol. 1995 Jan;13(1):8-10. doi: 10.1200/JCO.1995.13.1.8. No abstract available. PMID 7799047
- [Background] Pastorino U, Buyse M, Friedel G, Ginsberg RJ, Girard P, Goldstraw P, Johnston M, McCormack P, Pass H, Putnam JB Jr; International Registry of Lung Metastases. Long-term results of lung metastasectomy: prognostic analyses based on 5206 cases. J Thorac Cardiovasc Surg. 1997 Jan;113(1):37-49. doi: 10.1016/s0022-5223(97)70397-0. PMID 9011700
- [Background] Lievens Y, Guckenberger M, Gomez D, Hoyer M, Iyengar P, Kindts I, Mendez Romero A, Nevens D, Palma D, Park C, Ricardi U, Scorsetti M, Yu J, Woodward WA. Defining oligometastatic disease from a radiation oncology perspective: An ESTRO-ASTRO consensus document. Radiother Oncol. 2020 Jul;148:157-166. doi: 10.1016/j.radonc.2020.04.003. Epub 2020 Apr 22. PMID 32388150
- [Background] Lehrer EJ, Singh R, Wang M, Chinchilli VM, Trifiletti DM, Ost P, Siva S, Meng MB, Tchelebi L, Zaorsky NG. Safety and Survival Rates Associated With Ablative Stereotactic Radiotherapy for Patients With Oligometastatic Cancer: A Systematic Review and Meta-analysis. JAMA Oncol. 2021 Jan 1;7(1):92-106. doi: 10.1001/jamaoncol.2020.6146. PMID 33237270
- [Background] Zelefsky MJ, Yamada Y, Greco C, Lis E, Schoder H, Lobaugh S, Zhang Z, Braunstein S, Bilsky MH, Powell SN, Kolesnick R, Fuks Z. Phase 3 Multi-Center, Prospective, Randomized Trial Comparing Single-Dose 24 Gy Radiation Therapy to a 3-Fraction SBRT Regimen in the Treatment of Oligometastatic Cancer. Int J Radiat Oncol Biol Phys. 2021 Jul 1;110(3):672-679. doi: 10.1016/j.ijrobp.2021.01.004. Epub 2021 Jan 8. PMID 33422612
- [Background] Ryu S, Jin R, Jin JY, Chen Q, Rock J, Anderson J, Movsas B. Pain control by image-guided radiosurgery for solitary spinal metastasis. J Pain Symptom Manage. 2008 Mar;35(3):292-8. doi: 10.1016/j.jpainsymman.2007.04.020. Epub 2008 Jan 22. PMID 18215498
- [Background] Ryu S, Jin JY, Jin R, Rock J, Ajlouni M, Movsas B, Rosenblum M, Kim JH. Partial volume tolerance of the spinal cord and complications of single-dose radiosurgery. Cancer. 2007 Feb 1;109(3):628-36. doi: 10.1002/cncr.22442. PMID 17167762
- [Background] Zeng KL, Tseng CL, Soliman H, Weiss Y, Sahgal A, Myrehaug S. Stereotactic Body Radiotherapy (SBRT) for Oligometastatic Spine Metastases: An Overview. Front Oncol. 2019 May 1;9:337. doi: 10.3389/fonc.2019.00337. eCollection 2019. PMID 31119099
- [Background] Rusthoven KE, Kavanagh BD, Burri SH, Chen C, Cardenes H, Chidel MA, Pugh TJ, Kane M, Gaspar LE, Schefter TE. Multi-institutional phase I/II trial of stereotactic body radiation therapy for lung metastases. J Clin Oncol. 2009 Apr 1;27(10):1579-84. doi: 10.1200/JCO.2008.19.6386. Epub 2009 Mar 2. PMID 19255320
- [Background] Guckenberger M, Lievens Y, Bouma AB, Collette L, Dekker A, deSouza NM, Dingemans AC, Fournier B, Hurkmans C, Lecouvet FE, Meattini I, Mendez Romero A, Ricardi U, Russell NS, Schanne DH, Scorsetti M, Tombal B, Verellen D, Verfaillie C, Ost P. Characterisation and classification of oligometastatic disease: a European Society for Radiotherapy and Oncology and European Organisation for Research and Treatment of Cancer consensus recommendation. Lancet Oncol. 2020 Jan;21(1):e18-e28. doi: 10.1016/S1470-2045(19)30718-1. PMID 31908301
- [Background] Loi M, Alifano M, Scorsetti M, Nuyttens JJ, Livi L. Judging a Fish by Its Ability to Climb a Tree? A Call for Novel Endpoints in the Appraisal of Ablative Local Treatments of Oligometastatic Cancer. Oncologist. 2021 Jun;26(6):e1085-e1086. doi: 10.1002/onco.13747. Epub 2021 Apr 9. PMID 33686724
- [Background] Poon I, Erler D, Dagan R, Redmond KJ, Foote M, Badellino S, Biswas T, Louie AV, Lee Y, Atenafu EG, Ricardi U, Sahgal A. Evaluation of Definitive Stereotactic Body Radiotherapy and Outcomes in Adults With Extracranial Oligometastasis. JAMA Netw Open. 2020 Nov 2;3(11):e2026312. doi: 10.1001/jamanetworkopen.2020.26312. PMID 33196810
- [Background] Buglione M, Jereczek-Fossa BA, Bonu ML, Franceschini D, Fodor A, Zanetti IB, Gerardi MA, Borghetti P, Tomasini D, Di Muzio NG, Oneta O, Scorsetti M, Franzese C, Romanelli P, Catalano G, Dell'Oca I, Beltramo G, Ivaldi GB, Laudati A, Magrini SM, Antognoni P; Italian Society of Radiotherapy and Clinical Oncology - Regional Group Lombardy (AIROL). Radiosurgery and fractionated stereotactic radiotherapy in oligometastatic/oligoprogressive non-small cell lung cancer patients: Results of a multi-institutional series of 198 patients treated with "curative" intent. Lung Cancer. 2020 Mar;141:1-8. doi: 10.1016/j.lungcan.2019.12.019. Epub 2020 Jan 3. PMID 31926440
- [Background] Sindhu KK, Leiter A, Moshier E, Lin JY, Carroll E, Brooks D, Shimol JB, Eisenberg E, Gallagher EJ, Stock RG, Galsky MD, Buckstein M. Durable disease control with local treatment for oligoprogression of metastatic solid tumors treated with immune checkpoint blockade. Cancer Treat Res Commun. 2020;25:100216. doi: 10.1016/j.ctarc.2020.100216. Epub 2020 Oct 8. PMID 33049542
- [Background] Gaertner J, Elsner F, Pollmann-Dahmen K, Radbruch L, Sabatowski R. Electronic pain diary: a randomized crossover study. J Pain Symptom Manage. 2004 Sep;28(3):259-67. doi: 10.1016/j.jpainsymman.2003.12.017. PMID 15336338
- [Background] de Wit R, van Dam F, Hanneman M, Zandbelt L, van Buuren A, van der Heijden K, Leenhouts G, Loonstra S, Abu-Saad HH. Evaluation of the use of a pain diary in chronic cancer pain patients at home. Pain. 1999 Jan;79(1):89-99. doi: 10.1016/S0304-3959(98)00158-4. PMID 9928781
- [Background] Mizumoto M, Harada H, Asakura H, Hashimoto T, Furutani K, Hashii H, Takagi T, Katagiri H, Takahashi M, Nishimura T. Prognostic factors and a scoring system for survival after radiotherapy for metastases to the spinal column: a review of 544 patients at Shizuoka Cancer Center Hospital. Cancer. 2008 Nov 15;113(10):2816-22. doi: 10.1002/cncr.23888. PMID 18846565
- [Background] Cox BW, Spratt DE, Lovelock M, Bilsky MH, Lis E, Ryu S, Sheehan J, Gerszten PC, Chang E, Gibbs I, Soltys S, Sahgal A, Deasy J, Flickinger J, Quader M, Mindea S, Yamada Y. International Spine Radiosurgery Consortium consensus guidelines for target volume definition in spinal stereotactic radiosurgery. Int J Radiat Oncol Biol Phys. 2012 Aug 1;83(5):e597-605. doi: 10.1016/j.ijrobp.2012.03.009. Epub 2012 May 19. PMID 22608954
- [Background] Ryu S, Pugh SL, Gerszten PC, Yin FF, Timmerman RD, Hitchcock YJ, Movsas B, Kanner AA, Berk LB, Followill DS, Kachnic LA. RTOG 0631 phase 2/3 study of image guided stereotactic radiosurgery for localized (1-3) spine metastases: phase 2 results. Pract Radiat Oncol. 2014 Mar-Apr;4(2):76-81. doi: 10.1016/j.prro.2013.05.001. Epub 2013 Jun 4. PMID 24890347
- [Background] Timmerman RD. An overview of hypofractionation and introduction to this issue of seminars in radiation oncology. Semin Radiat Oncol. 2008 Oct;18(4):215-22. doi: 10.1016/j.semradonc.2008.04.001. No abstract available. PMID 18725106